CLINICAL TRIAL: NCT07122245
Title: Demographics of Lung Cancer in Female Patients: A Retrospective Based Analysis
Brief Title: Demographics of Lung Cancer in Females
Status: Recruiting | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Abd Elmoniem Mohamed, Lecturer of chest medicine faculty of medicine, Mansoura University Hospital
Other Study IDs: R.25.07.3275
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer
Keywords: Demographics; lung cancer; female patients
MeSH Terms: conditions — Lung Neoplasms | interventions — Demography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- bronchogenic carcinoma in female patients: A retrospective cohort study will be conducted on bronchogenic carcinoma female patients who had been presented to and diagnosed at chest diseases department, Oncology Center Mansoura University (OCMU).
  Interventions: Behavioral: Demographics and risk factors of lung cancer

INTERVENTIONS:
Behavioral: Demographics and risk factors of lung cancer — A retrospective cohort study will be conducted on bronchogenic carcinoma patients who had been presented to and diagnosed at chest diseases department, Oncology Center Mansoura University (OCMU).

SUMMARY:
Lung cancer has been the most common and fatal type of cancer; indeed worldwide incidence of lung cancer is alarming. It is considered a leading cause of cancer- related deaths among males and females due to environmental pollution, occupational exposure, genetic susceptibility, increasing number of smokers and others.

DETAILED DESCRIPTION:
Lung cancer has been the most common and fatal type of cancer; indeed worldwide incidence of lung cancer is alarming. It is considered a leading cause of cancer- related deaths among males and females due to environmental pollution, occupational exposure, genetic susceptibility, increasing number of smokers and others.

Moreover, a large proportion of people living in low and middle income countries are exposed to secondhand smoke (SHS) in their homes, workplaces, and other public places.

Although, lung cancer had become one of fatality causes of the 20th century due to an increasing life span combined with exposures to various etiologic factors, it is one of the leading causes of preventable deaths.

There are various important risk factors other than tobacco smoking that can contribute substantially to the lung cancer mortality in never smokers; these other lung carcinogens often act in an additive or synergistic manner in individuals who smoke tobacco products.

ELIGIBILITY:
Inclusion Criteria:

* All female patients presented with bronchogenic carcinoma patients and diagnosed at chest diseases department, Oncology Center Mansoura University (OCMU) in last 10 years.

Exclusion Criteria:

* lung metastasis ( not primary bronchogenic carcinoma)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — A retrospective cohort study will be conducted on bronchogenic carcinoma patients who had been presented to and diagnosed at chest diseases department, Oncology Center Mansoura University (OCMU) in last 10 years as smoking is a major risk factor and it is more common in males than females.
Study Population: A retrospective cohort study will be conducted on bronchogenic carcinoma patients who had been presented to and diagnosed at chest diseases department, Oncology Center Mansoura University (OCMU) in last 10 years.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2026-02-07 (Estimated); Study Completion 2026-04-07 (Estimated)

PRIMARY OUTCOMES:
Risk factors of lung cancer in females | 6 months
  A retrospective cohort study will be conducted on bronchogenic carcinoma patients who had been presented to and diagnosed at chest diseases department, Oncology Center Mansoura University (OCMU) in last 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AbdElmoniem, Principal Investigator — Lecturer of chest medicine faculty of medicine Mansoura university
Locations (1):
- Mohamed AbdElmoniem, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No